CLINICAL TRIAL: NCT05527977
Title: Pilot Demonstration for Physician Compensation Incentives to Improve Diagnostic Specificity in Clinical Documentation
Brief Title: Clinical Documentation Physician Compensation Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, David S. Burstein, Assistant Professor, Rush University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22060905-IRB01
Record Dates: First submitted 2022-08-26; First posted 2022-09-06 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Compensation Incentives; Clinical Documentation; Physician Work Environment; Diagnostic Error

STUDY DESIGN:
Intervention Model Description: To answer the research question, the investigators will extract data at the visit-level and perform the analysis at the physician-level. The investigators will perform descriptive statistics of physician and patient characteristics. Depending on the distribution of the data, the primary analysis will be paired t-test or Wilcoxon signed rank test comparing 6 weeks of baseline data for each physician to 12 weeks of data with compensation incentives. Performance by each physician during the baseline and incentivized periods will be assessed as a proportion at the visit level. The investigators will perform a multivariate interrupted time series as a sensitivity analysis. Patient and physician variables will be used as covariates in the multivariate analysis.
  The intevestigators will compare baseline documentation (Arm #1) with incentivized documentation (Arm #2)
Who Masked: Outcomes Assessor
Masking Description: The investigators have two research assistants who will perform retrospective chart review. The participants will not be informed of the incentive used (i.e., participants will now know whether the investigators have control/experimental group nor pre/post design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Period (No Intervention): Run-in non-incentivized period for all participants.
- Incentivized Period (Experimental): 3 month period during which time clinicians will receive compensation incentives for their performance in the program to improve clinical documentation.
  Interventions: Behavioral: Compensation Incentives to improve Clinical Documentation

INTERVENTIONS:
Behavioral: Compensation Incentives to improve Clinical Documentation — The investigators have identified six Diagnoses of Interest for the initiative. For each Diagnosis of Interest, the investigators have specified a series of clinically significant diagnostic details. Each physician will receive a compensation bonus from a pool of $20,000 based on the absolute number of times that he or she appropriately documented a Diagnosis of Interest.
  The investigators will use SQL Server Management Studio 18.0 to create an initial dataset using ICD-10 codes from office visits during which a Diagnosis of Interest was addressed. The investigators will compare documentation during the 12-week against a 6-week period prior to the intervention. The 6-week period will not be used to determine compensation bonuses. Two blinded research assistants will review H&P's and progress notes from extracted visits to tabulate the number of times that clinical documentation met expectations.
  Arms: Incentivized Period

SUMMARY:
Clinical documentation which omits significant medical details negatively affects communication among physicians and impedes the diagnostic process. Clinical documentation may be improved by using compensation incentives. Therefore, compensation incentives are a compelling mechanism to promote documentation of significant medical details to improve the diagnostic process.

The investigators' proposed project will use physician compensation incentives to improve documentation of clinically significant details for six common diagnoses in outpatient general internal medicine. The investigators will choose clinically significant details which more accurately represent patient complexity, improve the diagnostic process, and have potential to improve patient outcomes. To determine whether compensation incentives improve documentation of clinically significant details, the investigators will compare physicians' baseline documentation to incentivized documentation. The purpose of the investigators' project is to improve communication of clinically significant diagnostic information among physicians, thereby reducing suboptimal treatment plans, overuse, medical error, and cognitive burden upon physicians.

DETAILED DESCRIPTION:
Implementation: The investigators' proposed project will use physician compensation incentives to improve documentation of clinically significant details for six common diagnoses in outpatient general internal medicine. The purpose of the program is to improve clinical documentation in order to reduce misdiagnosis and medical errors. The investigators will invite 30-35 primary care physicians in internal medicine and family medicine within Rush University Medical Group to participate. The investigators will review participants' office visit notes for clinical documentation that meets pre-specified criteria. The investigators anticipate that physicians will receive a $5-$10 compensation bonus for each office visit progress note that meets clinical criteria. The investigators' program will be in effect for 3-months. The average performing physician is expected to receive $650-$700 in compensation incentives over the entire 3-month period (higher performing physicians expected to earn $1,000 or above for superior performance).

Approach: To determine whether compensation incentives improve documentation of clinically significant details, the investigators will compare physicians' baseline documentation (during a 6-week run-in period) to incentivized documentation (a 3-month period when physicians will receive compensation incentives for their clinical documentation). Two research assistants will perform retrospective chart review and audits of office visit progress notes. Notes will be scored for whether documentation includes pre-specified clinically significant information. For example, if a patient has had a Deep Vein Thrombosis (DVT), the investigators would assess whether the month of onset of the DVT and duration of anticoagulation therapy was documented in the note. The investigators anticipate that compensation incentives will improve physicians' clinical documentation of clinically significant medical details. The investigators' results will be reported in aggregate at the physician-level.

Participation: 30-35 physicians will be invited to participate in both the incentives program and analysis comparing baseline performance to incentivized performance. If a physician opts out of the analysis, that participant will not be eligible for compensation incentives. The investigators chose a sample of 30-35 physicians so that the study has enough power to detect a significant difference in performance in clinical documentation during the incentivized period compared to baseline.

Risks to patients: The investigators will use patient-level data as covariates in the analysis. The investigators' analysis will occur in a similar fashion as other retrospective studies, whereby patient-level information will be used from individual office visits in the analysis. Patient-level information will be de-identified as quickly as possible and precautions will be made to keep patient and physician-level data secure.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, PA's, and NP's at any of 8 pre-selected Rush practice sites.
* Clinical FTE >40%

Exclusion Criteria:

• Physicians, PA's, or NP's who have a significant change in clinical FTE or scheduled patient volume during the intervention

Equitable considerations include: Enrolling all clinicians (MD/DO, PA, NP) at each practice. Physicians with <40% FTE are expected to be eligible to earn low amounts of income from the program (estimated around less than $300 before taxes over 3-month period), hence the investigators will exclude them due to poor motivating force of this total incentive and adverse impacts on the statistical analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Documentation | Change from baseline documentation over 6 a week period to incentivized documentation over a 12 week period.
  2 Research assistants will use a binary scoring system for whether or not the documentation for a given diagnosis of interest includes pre-specified diagnostic information at the visit level. The investigators will create this binary scoring system a priori using evidence-based literature about common documentation errors and shortcomings related to the diagnostic process

CONTACTS AND LOCATIONS:
Overall Officials: David S Burstein, MD MS, Principal Investigator — Assistant Professor
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared only with the research team on record for the study.